CLINICAL TRIAL: NCT00003257
Title: A Phase II, Multicenter, Open Label Study to Evaluate Effectiveness and Safety of AdCMV-p53 Administered by Intra-Tumoral Injections in 39 Patients With Recurrent Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Gene Therapy in Treating Patients With Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aventis Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066148; AVENTIS-T-202; MCC-11653; RP-T-202; NCI-V98-1394
Record Dates: First submitted 1999-11-01; First posted 2004-09-10 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-04

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — advexin

INTERVENTIONS:
Biological: Ad5CMV-p53 gene

SUMMARY:
RATIONALE: Inserting the gene for p53 into a person's tumor may improve the body's ability to fight cancer or make the cancer more sensitive to chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of gene therapy in treating patients who have recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the objective response rate of Ad5CMV-p53 in patients with recurrent squamous cell carcinoma of the head and neck. II. Evaluate the duration of response, time to disease progression, and overall survival of these patients after this treatment. III. Evaluate the effectiveness of Ad5CMV-p53 in reducing cancer morbidity (pain assessment, analgesic consumption, and Karnofsky performance status). IV. Assess the quality of life of these patients receiving this treatment.

OUTLINE: This is a multicenter, open label study. All patients receive direct intratumoral injections of Ad5CMV-p53 on days 1, 2, and 3 of each 4-week treatment course. Patients are treated for at least 2 courses barring local disease progression or unacceptable adverse events; patients with responding or stable disease receive a maximum of 12 courses. Patients are evaluated for safety 4 weeks from the completion of the last treatment. Quality of life is assessed before, during, and after treatment. Patients are followed every 2 months for up to 18 months or until death.

PROJECTED ACCRUAL: A maximum of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck (SCCHN) Recurrent disease documented by histology or cytology (excluding endolaryngeal recurrence) following first line therapy with curative intent, such as: Radiation (at least 5000 cGy by standard methodology) and/or Surgery (definitive resection with postoperative radiation as indicated) Lesions accessible to intratumoral injections Bidimensionally measurable disease The sum of the products of the bidirectional measurements for all bidimensionally measurable lesions must be not greater than 30 cm2 The sum of the longest diameters of all measurable lesions must be not greater than 10 cm No CNS metastasis Tumor tissue from biopsy of primary or recurrent tumor must be available to determine p53 mutation status

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 2,000/mm3 Hepatic: Total bilirubin no greater than upper limit of normal (ULN) AST/SGOT and/or ALT/SGPT no greater than 1.5 times ULN Alkaline phosphatase no greater than 5 times ULN Renal: Not specified Other: Not pregnant or nursing Barrier contraception required during treatment Negative for HIV 1, HIV 2, hepatitis B, and hepatitis C At least 2 years since prior malignancy, other than SCCHN No contact with former tissue or organ transplant recipients or persons with severe immunodeficiency disease within 28 days following final dose of study drug No serious concurrent medical conditions No active uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunostimulating drugs No prior autologous or allogeneic organ or tissue transplant Chemotherapy: At least 4 weeks since prior chemotherapy At least 6 weeks since nitrosourea or mitomycin No other concurrent chemotherapy Endocrine therapy: No concurrent nontopical corticosteroids unless chronic (at least 6 months) at low doses (no greater than 10 mg of oral prednisone) Radiotherapy: See Disease Characteristics At least 4 weeks since radiotherapy to measurable disease sites, unless progressive disease No concurrent radiotherapy to disease sites receiving study drug injections Surgery: See Disease Characteristics No concurrent surgery to disease sites receiving study drug injections Other: No concurrent high dose steroids At least 4 weeks since experimental therapy No concurrent other experimental drugs or therapy No prior gene therapy using adenoviral vectors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Lyndah Dreiling, MD, Study Chair — Aventis Pharmaceuticals
Locations (10):
- United States (10):
  - Sidney Kimmel Cancer Center, San Diego, California
  - University of Colorado Cancer Center, Denver, Colorado
  - University of Connecticut School of Medicine, Farmington, Connecticut
  - Clinical Sciences Building, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Simmons Cancer Center - Dallas, Dallas, Texas